CLINICAL TRIAL: NCT05385198
Title: VOICE: Values, Opportunities, Integration, Control and Evaluation: Towards a Partnership Between Parents of Very Premature Infants and Healthcare Professionals in China
Brief Title: VOICE Study in China 'Towards a Partnership Between Parents of Very Premature Infants and Healthcare Professionals'
Acronym: VOICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HN06
Record Dates: First submitted 2022-04-30; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Emotional Stress; Parents; Family Separation; Neonatal Intensive Care; Parents Support; Family Centered Care; Infant ALL
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOICE care (Experimental): The VOICE conversations contain minimal 5 consecutive conversations with parents. The conversations are not rigid or strictly protocolized but rather focus on issues related to the situation of the admission period of the infant and the conversations should be individualized based on the parent needs. Thus, depending on the situation of the infant and the home situation of the parents.
  The content of the VOICE conversations is built up based on the admission pathway of the infant. Every VOICE conversation has its own focus, and these are presented in the 5 VOICE conversation guides. Basically, every VOICE conversation is about the support of parents and infant.
  The principles of the VOICE conversations are Values, Opportunities, Integration, Control and Evaluation. The VOICE program focuses on a systematic and planned communications with parents during the NICU admission and follow-up 2-4 weeks after NICU discharge.
  Interventions: Behavioral: VOICE care
- Standard care (No Intervention): Standard care is defined as the standard family centered care (FCC) practices currently implemented in the NICU. Parents are allowed to visit the NICU for 3 hours every day and provide basic care to their infant. Standard care involves meetings with the doctors three times a week and the content is mainly directed to the medical condition and treatments of the infant. No other meetings between parents and doctors/nurses exists. The FCC principles implicate that parents and NICU staff work closely together on the NICU. This also involves unscheduled information and communication contact moments where short questions of parents will be addressed.

INTERVENTIONS:
Behavioral: VOICE care — I phase:build a relationship with parents and where the Values of the parents and NICU staff is shared.
  II phase: discuss with the parents the Opportunities the parents can have to be more involved in the care of their baby.
  III phase: Integration of the involvement of the parents in the care of their baby. The experiences of parents need to be shared with the NICU staff. Any raising issue about the involvement of care by the parents can be discussed and see if improvement is needed.
  IV phase:Control of the knowledge about the care of their baby before going home and if the parents have any issues which need to be arranged before discharge.
  V phase:Evaluation. During this conversation the overall experiences of the parents will be discussed and if there are any further questions related to the care of their baby at home will be explored and discussed.
  Arms: VOICE care

SUMMARY:
Background: Admission to a Neonatal Intensive Care Unit (NICU) is associated with significant levels of parental stress and anxiety. Parents are often uncertain to perform care giving activities and might feel uncertain to fulfill the desirable parental role during NICU admission. Furthermore, transition of the NICU to another unit or hospital is stressful for parents often related to poor information and communication. A VOICE program is developed aiming to increase the empowerment of parents, to improve partnership between parents of very premature infants and healthcare professionals.

Aim: To conduct a feasibility RCT study to evaluate the implementation and the effect of the VOICE program on parental stress and anxiety in the NICU.

Methods:

Design is a feasibility RCT to test the procedures, compliance, determine sample size, estimating recruitment and retention, and to get first insight in the effects of the VOICE program on the outcome measures.

VOICE will be implemented as a structured empowerment and partnership program for parents from admission of the infant to the NICU till the first visit to the out-patient clinic. The program exists of five structured and focused meetings, following the acronym VOICE (Values, Opportunities, Integration, Control and Evaluation). These interdisciplinary meetings with parents aim to increase the involvement of parents in the care and decision making of participants' infant in the NICU. The primary outcome measures will be parental stress and anxiety measured by the Chinese version of the Hospital Anxiety and Depression scale (HADS) and the Edinburgh Postnatal Depression Scale (Chinese version). The secondary outcome measures will be parent satisfaction with care measured by the Empowerment of Parents in the Intensive Care (EMPATHIC-30) scale, length-of-stay in the NICU, hours of parental visitation and activities, compliance of NICU staff to the VOICE program.

An embedded qualitative study will be designed to explore the experiences of parents and NICU staff about the implemented VOICE program. Individual interviews with parents and focus groups sessions with NICU staff will be conduction. This will help to identify methodological issues such as recruitment and retention and any enablers and barriers to the intervention which may impede the future RCT.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONAL Preterm birth and admission at the Neonatal Intensive Care Unit (NICU) can be stressful and traumatic events both for parents and infants.

Infants born very premature are usually admitted to a NICU. A multidisciplinary dedicated team takes care of these infants and parents. Admission to a NICU is essential if the infant requires additional life support for their vital functions after birth. NICU admission is associated with high rates of impaired development of the infants, and parents or families often experience significant disruption, stress and anxiety during NICU admission and beyond.

Depending the diagnostic criteria, 6.8-16.5% of the mothers suffers of post-partum depression. Elevated stress levels and depressive symptoms are present upon NICU admission. Besides the normal stress of parenthood, parental distress is related to different factors such as physical and emotional isolation from the infant, a lack of control, adapting the idea of having a sick infant and the stress of the NICU environment.

During admission, support of nurses and doctors is important; when perception of nursing support is decreasing, mothers' depressive symptoms are increasing. Stress is known to negatively influence the parent-child relationship. Schappin concluded that stress decreases by better quality of care and stress in parents of premature infants is higher in comparison with term infants. Counseling parents in taking care of their infants is therefore very important.

The quality of care in the first weeks has a impact on parental stress. For optimal development of the infant, parents need to be involved in the total care process at the NICU. Creating an environment, both physical and emotional, in which involvement of parents is crucial in the care for their infant, increases outcome and decreases parental stress. In addition, maternal visits are positive associated with decreased length-of-stay and rates of behavioral and emotional problems. The main predictors of lower maternal NICU visitation were the number of potential traumatic events, maternal anxiety and number of children at home.

A program was developed called VOICE: Values, Opportunities, Integration, Control and Evaluation. The program exists of 5 structured meetings in congruence with the acronym VOICE: structural interdisciplinary meetings with parents to inform and communicate with parents and to support them in decision-making and care of their infant. The aim of this VOICE program is to decrease the level of parental stress in parents. To increase the parental involvement in decision-making and care, investigators aim to implement the VOICE program and test its feasibility and impact on parents.

AIM AND OBJECTIVES The aim of the feasibility RCT is to evaluate the implementation and the effect of the VOICE program on parental stress and anxiety in the NICU.

Specifically, the objectives are:

1. To determine the feasibility of delivering the VOICE program intervention to parents of infants GA <32 weeks admitted to the NICU A feasibility study will be conducted to collect process, resource, management and scientific data to inform the design of a larger multi-center RCT. The proposed outcome measures will be related to stress, anxiety, parent satisfaction, NICU length-of-stay, hours of parental visitation and their activities, compliance of NICU staff to the VOICE program.
2. To explore the implementation of the VOICE program intervention with parents and healthcare professionals.

A qualitative study will explore experiences of parents who will be participating in the feasibility study and the NICU staff carrying out the intervention. This will provide information on methodological issues such as recruitment/retention, and enablers/barriers of the intervention.

METHODS Design Design of the study is a feasibility study. Since the VOICE program is a complex intervention, the MRC-framework for developing and testing complex interventions will be followed. The process from development through to implementation of a complex intervention may take a wide range of different forms.

In the developmental phase, the VOICE intervention was developed from the available evidence and experts in this field, including parents. All involved healthcare professionals have been trained. After the developmental phase, the current 'step' in this MRC framework is the feasibility and piloting phase. The study will be a mixed-method study. Specifically, the feasibility study will be conducted with RCT design and an embedded qualitative design.

Setting The NICU of the Hunan Children's Hospital is a tertiary neonatal center providing high quality care and treatment. Infants above 24 weeks gestational age (GA) are admitted and treated in this NICU. More than 5000 newborns are admitted annually. Of these infants, around 350 are born very premature, with a GA <32 weeks. These very premature infants need long-term intensive care treatment with a mean length-of-stay of 35 days. The NICU has meanwhile implemented successfully family-centered care and parent are allowed to visit their infants and become more involved in the care.

Sample size As this is a feasibility study the sample size has been determined pragmatically to address the study objectives. Investigators aim to include parents (father and/or mother) of 30 infants in the intervention group and parents of 30 infants in the standard care group.

ELIGIBILITY:
Inclusion Criteria:

* Parents of infants born < 32 weeks GA
* Parents of infants admitted to NICU within 7days after birth
* Parents speaking and writing Chinese.

Exclusion Criteria:

* Parent of infants with an expected NICU length-of-stay less than 4 weeks
* Parents of infants having a major life-threatening congenital anomaly
* Parents of infants with a critical illness and unlikely to survive
* Parents with an inability to participate (health, family, social, or language issues that might inhibit their ability to collaborate with the NICU staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Hospital Anxiety and Depression before and after intervention | Time Frame of measurement : T1 = Baseline pre-intervention (first week of admission) , T2 = After intervention (4 weeks after discharge)
  Hospital Anxiety and Depression scale is a 14-item scale measuring hospital anxiety and depression. Seven of the items relate to anxiety and seven relate to depression. Each subscale has a score ranging from 0 to 21. Items are rated on a 4-point Likert scale, ranging from 0-3, generating a scale range of 0-42 points, with higher scores representing greater symptom severity. Score of 0-7 indicates normal levels of anxiety and depression; 8-10 indicate borderline abnormal anxiety and depression levels, and 11-21 suggest abnormal levels of anxiety and depression.

SECONDARY OUTCOMES:
Postnatal Depression | Measure time point: After invervention(4 weeks after discharge)
  Edinburgh Postnatal Depression Scale usually be completed in less than 5 minutes. Responses are scored 0, 1, 2, or 3 according to increased severity of the symptom. The total score is determined by adding together the scores for each of the 10 items. Cut-off scores ranged from 9 to 13 points and with higher scores representing greater symptom severity.
Parent satisfaction | Measure time point: After invervention(4 weeks after discharge)
  Parent satisfaction measured by the Empowerment of Parents in the Intensive Care (EMPATHIC-30) scale.The EMPATHIC-30 consist of 30 statement measuring parent satisfaction and experience. The scores of the statement are on a scale of 1-6 (from certainly yes to certainly no). Scores are presented in mean and SD values on statement level and domain level. Higher scores represent greater satisfaction.
Length-of-stay in the NICU | Measure time point: After invervention(4 weeks after discharge)
  The length-of-stay in the NICU will be collected.
Hours of parental daily visitation and their activities | Daily during intervention
  The number of hours of parental visitation and their activities will be collected.
Weight gain during hospitalization | T1 = at admission ,T2 = at discharge
  Weight at admission and weight at discharge will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-ming Peng, Principal Investigator — Hunan Children's Hospital

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Alkozei A, McMahon E, Lahav A. Stress levels and depressive symptoms in NICU mothers in the early postpartum period. J Matern Fetal Neonatal Med. 2014 Nov;27(17):1738-43. doi: 10.3109/14767058.2014.942626. Epub 2014 Jul 30. PMID 25005861
- [Background] Ayers S, Joseph S, McKenzie-McHarg K, Slade P, Wijma K. Post-traumatic stress disorder following childbirth: current issues and recommendations for future research. J Psychosom Obstet Gynaecol. 2008 Dec;29(4):240-50. doi: 10.1080/01674820802034631. PMID 18608815
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Davis L, Edwards H, Mohay H, Wollin J. The impact of very premature birth on the psychological health of mothers. Early Hum Dev. 2003 Aug;73(1-2):61-70. doi: 10.1016/s0378-3782(03)00073-2. PMID 12932894
- [Background] Engelhard IM, van den Hout MA, Schouten EG. Neuroticism and low educational level predict the risk of posttraumatic stress disorder in women after miscarriage or stillbirth. Gen Hosp Psychiatry. 2006 Sep-Oct;28(5):414-7. doi: 10.1016/j.genhosppsych.2006.07.001. PMID 16950377
- [Background] Engelhard IM, van Rij M, Boullart I, Ekhart TH, Spaanderman ME, van den Hout MA, Peeters LL. Posttraumatic stress disorder after pre-eclampsia: an exploratory study. Gen Hosp Psychiatry. 2002 Jul-Aug;24(4):260-4. doi: 10.1016/s0163-8343(02)00189-5. PMID 12100837
- [Background] Gonya J, Martin E, McClead R, Nelin L, Shepherd E. Empowerment programme for parents of extremely premature infants significantly reduced length of stay and readmission rates. Acta Paediatr. 2014 Jul;103(7):727-31. doi: 10.1111/apa.12669. PMID 24766486
- [Background] Greene MM, Rossman B, Patra K, Kratovil A, Khan S, Meier PP. Maternal psychological distress and visitation to the neonatal intensive care unit. Acta Paediatr. 2015 Jul;104(7):e306-13. doi: 10.1111/apa.12975. Epub 2015 Feb 27. PMID 25684177
- [Background] Helder OK, Verweij JC, van Staa A. Transition from neonatal intensive care unit to special care nurseries: experiences of parents and nurses. Pediatr Crit Care Med. 2012 May;13(3):305-11. doi: 10.1097/PCC.0b013e3182257a39. PMID 21705956
- [Background] Jiang S, Warre R, Qiu X, O'Brien K, Lee SK. Parents as practitioners in preterm care. Early Hum Dev. 2014 Nov;90(11):781-5. doi: 10.1016/j.earlhumdev.2014.08.019. Epub 2014 Sep 20. PMID 25246323
- [Background] Koren, P. E., DeChillo, N., & Friesen, B. J. (1992). Measuring empowerment in families whose children have emotional disabilities: A brief questionnaire. Rehabilitation Psychology, 37(4), 305-321.
- [Background] Latour JM, Duivenvoorden HJ, Hazelzet JA, van Goudoever JB. Development and validation of a neonatal intensive care parent satisfaction instrument. Pediatr Crit Care Med. 2012 Sep;13(5):554-9. doi: 10.1097/PCC.0b013e318238b80a. PMID 22460771
- [Background] Latour JM, Hazelzet JA, Duivenvoorden HJ, van Goudoever JB. Perceptions of parents, nurses, and physicians on neonatal intensive care practices. J Pediatr. 2010 Aug;157(2):215-220.e3. doi: 10.1016/j.jpeds.2010.02.009. Epub 2010 Mar 31. PMID 20359714
- [Background] Melnyk BM, Feinstein NF. Reducing hospital expenditures with the COPE (Creating Opportunities for Parent Empowerment) program for parents and premature infants: an analysis of direct healthcare neonatal intensive care unit costs and savings. Nurs Adm Q. 2009 Jan-Mar;33(1):32-7. doi: 10.1097/01.NAQ.0000343346.47795.13. PMID 19092521
- [Background] O'Brien K, Bracht M, Robson K, Ye XY, Mirea L, Cruz M, Ng E, Monterrosa L, Soraisham A, Alvaro R, Narvey M, Da Silva O, Lui K, Tarnow-Mordi W, Lee SK. Evaluation of the Family Integrated Care model of neonatal intensive care: a cluster randomized controlled trial in Canada and Australia. BMC Pediatr. 2015 Dec 15;15:210. doi: 10.1186/s12887-015-0527-0. PMID 26671340
- [Background] Schappin R, Wijnroks L, Uniken Venema MM, Jongmans MJ. Rethinking stress in parents of preterm infants: a meta-analysis. PLoS One. 2013;8(2):e54992. doi: 10.1371/journal.pone.0054992. Epub 2013 Feb 6. PMID 23405105
- [Background] Stowe ZN, Nemeroff CB. Women at risk for postpartum-onset major depression. Am J Obstet Gynecol. 1995 Aug;173(2):639-45. doi: 10.1016/0002-9378(95)90296-1. PMID 7645646
- [Background] Weis J, Zoffmann V, Egerod I. Improved nurse-parent communication in neonatal intensive care unit: evaluation and adjustment of an implementation strategy. J Clin Nurs. 2014 Dec;23(23-24):3478-89. doi: 10.1111/jocn.12599. Epub 2014 Apr 3. PMID 24698260
- [Background] White T , Matthey S , Boyd K , et al. Postnatal depression and post-traumatic stress after childbirth: Prevalence, course and co-occurrence[J]. Journal of Reproductive & Infant Psychology, 2006, 24(2):107-120.
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879